CLINICAL TRIAL: NCT02378285
Title: Treatment of Epicondylitis by Ultrasound-guided Local Injections of Autologous Conditioned Plasma (ACP®): a Double-blind Placebo-controlled Randomized Clinical Trial With One-year Follow-up
Brief Title: Treatment of Epicondylitis by Ultrasound-guided Local Injections of PRP (Platelet Rich Plasma)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arthrex SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ArthrexFR-001; 2009-A00804-53 (Other: ANSM)
Record Dates: First submitted 2015-02-23; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Epicondylitis
Keywords: recent lateral humeral epicondylitis; platelet-rich plasma; infiltration; tennis elbow; ultrasonography
MeSH Terms: conditions — Tennis Elbow | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP group (Active Comparator): ACP infiltration: 2 mL at 0 and 4 weeks with ultrasound guidance
  Interventions: Device: ACP
- Saline solution group (Placebo Comparator): Saline solution infiltration: 2mL at 0 and 4 weeks with ultrasound guidance
  Interventions: Other: Saline solution

INTERVENTIONS:
Device: ACP — ACP is prepared using the Autologous Conditioned Plasma (ACP®) device from Arthrex (Naples, Florida, USA), following the supplier instructions. 2 mL of ACP are transferred in a standard 2 mL injection syringe by a nurse. The standard 2 mL injection syringe is then given to the physician.The patient is installed on a table with his arm in supine position. A local subcutaneous anesthesia (2 ml of 1% lidocaine) is done just before the infiltration by the physician. The infiltration is then done guided by ultrasound.
  Arms: PRP group
Other: Saline solution — 2 mL of saline solution are placed in a standard injection syringe by a nurse. The syringe is then given to the physician. The patient is installed on a table with his arm in supine position. A local subcutaneous anesthesia (2 ml of 1% lidocaine) is done just before the infiltration by the physician. The infiltration is then done guided by ultrasound.
  Arms: Saline solution group

SUMMARY:
The purpose of this study is to assess efficacy of two intra-tendinous injections of platelet-rich plasma (PRP) on epicondylitis of recent evolution (≤ 3 months) compared compared to two intra-tendinous injections of saline solution (placebo).

DETAILED DESCRIPTION:
This was a prospective double-blind placebo-controlled randomized trial. Two ultrasound-guided injections of either PRP (ACP®, Arthrex) or saline solution were performed at 4 weeks interval.

Exclusion criterion was previous corticosteroid infiltration. All infiltrations were performed by Dr Bernard Montalvan. The selection of patients and the evaluation were conducted by Dr Patrick Le Goux who did not know which treatment had been allocated to which patient.

In the facility, no one apart from the investigators had access to full patient data.

An independent company represented by Mrs Amandine Ramseyer was hired to design, follow and carry the statistical analysis of the study. The data she got from the investigators were anonymous.

Patients were monitored by an independent evaluator blinded to treatment at baseline and 1, 3, 6 and 12 months follow-up.

Secondary criteria were the Roles-Maudsley score and the assessment of pain on isometric contraction of the extensor carpi radialis brevis and of the extensor digitorum communis.

The main evaluation criterion was the relative improvement from baseline to 6 months in pain score on visual analog scale (0-10).

Intragroup and intergroup intention-to-treat analyses were performed using Student's t-tests, applying the last-observation carried forward method. Differences of proportions were tested using chi-square. The sample size calculated was 22 patients per group so that this study had a power of 90% with typeI error rate α=0.05 to demonstrate a significant greater improvement of the global pain score of at least 10%, in the PRP over the placebo group with a standard deviation of 0.10. A "p" value of less than 0.05 was considered to be statistically significant. The SPSS software (version 19 for Windows) was used to perform statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from tennis elbow for less than three months
* Patients having never received former medical or orthopedic treatment for tennis elbow

Exclusion Criteria:

* Patients having received any treatment for this specific pathology
* Evidence of ongoing tumoral affection (controlled by MRI)
* Tennis elbow history
* Elbow fracture history
* Associated elbow pathology
* Inflammatory rheumatic disorders
* Bleeding disorders
* Ongoing anticoagulation therapy
* Allergy to local anesthetic
* Ongoing or previous cancer affection
* Pregnancy
* Diabetes

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Global pain score | 1 year

SECONDARY OUTCOMES:
Roles and Maudsley score | 1 year
Pain on ECRB* contraction | 1 year
  % positive
Pain on EDC** contraction | 1 year
  % positive

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Hardy, Pr, Study Director — Hospital Ambroise Paré Paris
Locations (1):
- Hôpital Ambroise Paré, Boulogne, France

REFERENCES:
- [Background] De Smedt T, de Jong A, Van Leemput W, Lieven D, Van Glabbeek F. Lateral epicondylitis in tennis: update on aetiology, biomechanics and treatment. Br J Sports Med. 2007 Nov;41(11):816-9. doi: 10.1136/bjsm.2007.036723. Epub 2007 Jul 6. PMID 17616547
- [Background] Nirschl RP. Elbow tendinosis/tennis elbow. Clin Sports Med. 1992 Oct;11(4):851-70. PMID 1423702
- [Background] McCormack RR Jr, Inman RD, Wells A, Berntsen C, Imbus HR. Prevalence of tendinitis and related disorders of the upper extremity in a manufacturing workforce. J Rheumatol. 1990 Jul;17(7):958-64. PMID 2213764
- [Background] Ono Y, Nakamura R, Shimaoka M, Hiruta S, Hattori Y, Ichihara G, Kamijima M, Takeuchi Y. Epicondylitis among cooks in nursery schools. Occup Environ Med. 1998 Mar;55(3):172-9. doi: 10.1136/oem.55.3.172. PMID 9624268
- [Background] Shiri R, Viikari-Juntura E. Lateral and medial epicondylitis: role of occupational factors. Best Pract Res Clin Rheumatol. 2011 Feb;25(1):43-57. doi: 10.1016/j.berh.2011.01.013. PMID 21663849
- [Background] Hamilton PG. The prevalence of humeral epicondylitis: a survey in general practice. J R Coll Gen Pract. 1986 Oct;36(291):464-5. PMID 3440991
- [Background] Murtagh JE. Tennis elbow. Aust Fam Physician. 1988 Feb;17(2):90-1, 94-5. No abstract available. PMID 3358752
- [Background] Smidt N, Lewis M, Hay EM, Van der Windt DA, Bouter LM, Croft P. A comparison of two primary care trials on tennis elbow: issues of external validity. Ann Rheum Dis. 2005 Oct;64(10):1406-9. doi: 10.1136/ard.2004.029363. Epub 2005 Mar 30. PMID 15800009
- [Background] Bisset L, Beller E, Jull G, Brooks P, Darnell R, Vicenzino B. Mobilisation with movement and exercise, corticosteroid injection, or wait and see for tennis elbow: randomised trial. BMJ. 2006 Nov 4;333(7575):939. doi: 10.1136/bmj.38961.584653.AE. Epub 2006 Sep 29. PMID 17012266
- [Background] Lindenhovius A, Henket M, Gilligan BP, Lozano-Calderon S, Jupiter JB, Ring D. Injection of dexamethasone versus placebo for lateral elbow pain: a prospective, double-blind, randomized clinical trial. J Hand Surg Am. 2008 Jul-Aug;33(6):909-19. doi: 10.1016/j.jhsa.2008.02.004. PMID 18656765
- [Background] Newcomer KL, Laskowski ER, Idank DM, McLean TJ, Egan KS. Corticosteroid injection in early treatment of lateral epicondylitis. Clin J Sport Med. 2001 Oct;11(4):214-22. doi: 10.1097/00042752-200110000-00002. PMID 11753057
- [Background] Roukis TS, Zgonis T, Tiernan B. Autologous platelet-rich plasma for wound and osseous healing: a review of the literature and commercially available products. Adv Ther. 2006 Mar-Apr;23(2):218-37. doi: 10.1007/BF02850128. PMID 16751155
- [Background] Ranly DM, McMillan J, Keller T, Lohmann CH, Meunch T, Cochran DL, Schwartz Z, Boyan BD. Platelet-derived growth factor inhibits demineralized bone matrix-induced intramuscular cartilage and bone formation. A study of immunocompromised mice. J Bone Joint Surg Am. 2005 Sep;87(9):2052-64. doi: 10.2106/JBJS.D.02752. PMID 16140821
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Borzini P, Mazzucco L. Tissue regeneration and in loco administration of platelet derivatives: clinical outcome, heterogeneous products, and heterogeneity of the effector mechanisms. Transfusion. 2005 Nov;45(11):1759-67. doi: 10.1111/j.1537-2995.2005.00600.x. PMID 16271101
- [Background] de Mos M, van der Windt AE, Jahr H, van Schie HT, Weinans H, Verhaar JA, van Osch GJ. Can platelet-rich plasma enhance tendon repair? A cell culture study. Am J Sports Med. 2008 Jun;36(6):1171-8. doi: 10.1177/0363546508314430. Epub 2008 Mar 7. PMID 18326832
- [Background] Foster TE, Puskas BL, Mandelbaum BR, Gerhardt MB, Rodeo SA. Platelet-rich plasma: from basic science to clinical applications. Am J Sports Med. 2009 Nov;37(11):2259-72. doi: 10.1177/0363546509349921. PMID 19875361
- [Background] Mazzocca AD, McCarthy MB, Chowaniec DM, Cote MP, Romeo AA, Bradley JP, Arciero RA, Beitzel K. Platelet-rich plasma differs according to preparation method and human variability. J Bone Joint Surg Am. 2012 Feb 15;94(4):308-16. doi: 10.2106/JBJS.K.00430. PMID 22336969
- [Background] Mishra AK, Skrepnik NV, Edwards SG, Jones GL, Sampson S, Vermillion DA, Ramsey ML, Karli DC, Rettig AC. Efficacy of platelet-rich plasma for chronic tennis elbow: a double-blind, prospective, multicenter, randomized controlled trial of 230 patients. Am J Sports Med. 2014 Feb;42(2):463-71. doi: 10.1177/0363546513494359. Epub 2013 Jul 3. PMID 23825183
- [Background] Creaney L, Wallace A, Curtis M, Connell D. Growth factor-based therapies provide additional benefit beyond physical therapy in resistant elbow tendinopathy: a prospective, single-blind, randomised trial of autologous blood injections versus platelet-rich plasma injections. Br J Sports Med. 2011 Sep;45(12):966-71. doi: 10.1136/bjsm.2010.082503. Epub 2011 Mar 15. PMID 21406450
- [Background] Thanasas C, Papadimitriou G, Charalambidis C, Paraskevopoulos I, Papanikolaou A. Platelet-rich plasma versus autologous whole blood for the treatment of chronic lateral elbow epicondylitis: a randomized controlled clinical trial. Am J Sports Med. 2011 Oct;39(10):2130-4. doi: 10.1177/0363546511417113. Epub 2011 Aug 2. PMID 21813443
- [Background] Raeissadat SA, Sedighipour L, Rayegani SM, Bahrami MH, Bayat M, Rahimi R. Effect of Platelet-Rich Plasma (PRP) versus Autologous Whole Blood on Pain and Function Improvement in Tennis Elbow: A Randomized Clinical Trial. Pain Res Treat. 2014;2014:191525. doi: 10.1155/2014/191525. Epub 2014 Jan 20. PMID 24579044
- [Background] Giusti I, Rughetti A, D'Ascenzo S, Millimaggi D, Pavan A, Dell'Orso L, Dolo V. Identification of an optimal concentration of platelet gel for promoting angiogenesis in human endothelial cells. Transfusion. 2009 Apr;49(4):771-8. doi: 10.1111/j.1537-2995.2008.02033.x. Epub 2008 Dec 23. PMID 19170984
- [Background] de Vos RJ, Windt J, Weir A. Strong evidence against platelet-rich plasma injections for chronic lateral epicondylar tendinopathy: a systematic review. Br J Sports Med. 2014 Jun;48(12):952-6. doi: 10.1136/bjsports-2013-093281. Epub 2014 Feb 21. PMID 24563387
- [Derived] Montalvan B, Le Goux P, Klouche S, Borgel D, Hardy P, Breban M. Inefficacy of ultrasound-guided local injections of autologous conditioned plasma for recent epicondylitis: results of a double-blind placebo-controlled randomized clinical trial with one-year follow-up. Rheumatology (Oxford). 2016 Feb;55(2):279-85. doi: 10.1093/rheumatology/kev326. Epub 2015 Sep 8. PMID 26350485